CLINICAL TRIAL: NCT02274766
Title: ADS-5102 (Amantadine HCl) Extended Release Efficacy and Safety Study in Parkinson's Disease Patients With Levodopa-Induced Dyskinesia (EASE LID 3 Study)
Brief Title: Efficacy and Safety Study of ADS-5102 in PD Patients With Levodopa-Induced Dyskinesia
Acronym: EASE LID 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Adamas Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADS-AMT-PD304
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Results first posted 2018-01-10 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Dyskinesia; Levodopa-Induced Dyskinesia (LID); Parkinson's Disease (PD)
Keywords: Levodopa-Induced Dyskinesia; LID; Parkinsonism; Parkinson's Disease
MeSH Terms: conditions — Dyskinesias; Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADS-5102 (amantadine HCl extended release) (Experimental): ADS-5102 (amantadine HCl extended release)
  Interventions: Drug: ADS-5102
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ADS-5102 — Oral capsules to be administered once nightly at bedtime, for 13 weeks.
  Other Names: amantadine HCl extended release
  Arms: ADS-5102 (amantadine HCl extended release)
Other: Placebo — Oral capsules to be administered once nightly at bedtime, for 13 weeks.
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled, 2-arm, parallel group study to evaluate the efficacy and safety of ADS-5102 extended release (ER) capsules, an investigational formulation of amantadine, dosed once nightly at bedtime for the treatment of levodopa-induced dyskinesia (LID) in subjects with Parkinson's disease (PD). The novel pharmacokinetic profile of ADS-5102 is expected to achieve i) maximal concentrations in the early morning through mid-day, when LID can be troublesome, and ii) lower concentrations in the evening, potentially reducing the negative impact of amantadine on sleep. This pharmacokinetic profile could enable higher doses to be tolerated with a once-nightly ER formulation than can be tolerated with an immediate-release formulation. The once-nightly dosing regimen may also provide enhanced convenience and compliance.

In a previous clinical study, ADS-5102 met its primary endpoint; LID was significantly reduced as measured by the change in UDysRS score over 8 weeks vs. placebo.

ELIGIBILITY:
Inclusion Criteria:

* Signed a current IRB/REB/IEC-approved informed consent form;
* Parkinson's disease, per UK Parkinson's Disease Society (UKPDS) Brain Bank Clinical Diagnostic Criteria;
* On a stable regimen of antiparkinson's medications for at least 30 days prior to screening, including a levodopa preparation administered not less than three times daily, and willing to continue the same doses and regimens during study participation;
* Following diary training, the subject is willing and able to understand and complete the 24-hour PD home diary (trained caregiver/study partner assistance allowed);
* Any other current and allowed prescription/non-prescription medications and/or nutritional supplements taken regularly must have been at a stable dose and regimen for at least 30 days prior to screening, and subject must be willing to continue the same doses and regimens during study participation (this criterion does not apply to medications that are being taken pre-study only on an as-needed basis);

Exclusion Criteria:

* History of neurosurgical intervention related to Parkinson's disease (e.g. deep brain stimulation);
* History of seizures within 2 years prior to screening;
* History of stroke or TIA within 2 years prior to screening;
* History of cancer within 5 years prior to screening, with the following exceptions: adequately treated non-melanomatous skin cancers, localized bladder cancer, non-metastatic prostate cancer, in situ cervical cancer, or other definitively treated cancer that is considered cured;
* Presence of cognitive impairment, as evidenced by a Mini-Mental Status Examination (MMSE) score of less than 24 during screening;
* If female, is pregnant or lactating;
* If a sexually active female, is not surgically sterile or at least 2 years post-menopausal, or does not agree to utilize an effective method of contraception from screening through at least 4 weeks after the completion of study treatment, using one of the following: barrier methods (diaphragm or partner using condoms plus use of spermicidal jelly or foam, preferably double-barrier methods); oral or implanted hormonal contraceptive; intrauterine device (IUD); or vasectomized male partner;
* Treatment with an investigational drug or device within 30 days prior to screening;
* Treatment with an investigational biologic within 6 months prior to screening;
* Current participation in another clinical trial;

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03-10 (Actual); Study Completion 2016-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials Director, Study Director — Adamas Pharmaceuticals, Inc.
Locations (45):
- United States (21):
  - Fountain Valley, California
  - Sunnyvale, California
  - Boca Raton, Florida
  - Jacksonville, Florida
  - Port Charlotte, Florida
  - Sunrise, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Kansas City, Kansas
  - Baltimore, Maryland
  - Elkridge, Maryland
  - Boston, Massachusetts
  - West Bloomfield, Michigan
  - Greensboro, North Carolina
  - Raleigh, North Carolina
  - Tulsa, Oklahoma
  - Roanoke, Virginia
  - Kirkland, Washington
  - Morgantown, West Virginia
  - Milwaukee, Wisconsin
- Austria (2):
  - Innsbruck
  - Vienna
- France (11):
  - Bordeaux
  - Bron
  - Clermont-Ferrand
  - Lille
  - Marseille
  - Montpellier
  - Poitier
  - Rennes
  - Rouen
  - Strasbourg
  - Toulouse
- Germany (10):
  - München, Bavaria
  - Beelitz-Heilstätten, Brandenburg
  - Göttingen, Lower Saxony
  - Leipzig, Saxony
  - Gera, Thuringia
  - Stadtroda, Thuringia
  - Berlin
  - Hamburg
  - Kassel
  - Marburg
- Barcelona, Spain

REFERENCES:
- [Derived] Hauser RA, Mehta SH, Kremens D, Chernick D, Formella AE. Effects of Gocovri (Amantadine) Extended-Release Capsules on Motor Aspects of Experiences of Daily Living in People with Parkinson's Disease and Dyskinesia. Neurol Ther. 2021 Dec;10(2):739-751. doi: 10.1007/s40120-021-00256-1. Epub 2021 May 22. PMID 34024025
- [Derived] Mehta SH, Pahwa R, Tanner CM, Hauser RA, Johnson R. Effects of Gocovri (Amantadine) Extended Release Capsules on Non-Motor Symptoms in Patients with Parkinson's Disease and Dyskinesia. Neurol Ther. 2021 Jun;10(1):307-320. doi: 10.1007/s40120-021-00246-3. Epub 2021 Apr 17. PMID 33864229
- [Derived] Elmer LW, Juncos JL, Singer C, Truong DD, Criswell SR, Parashos S, Felt L, Johnson R, Patni R. Pooled Analyses of Phase III Studies of ADS-5102 (Amantadine) Extended-Release Capsules for Dyskinesia in Parkinson's Disease. CNS Drugs. 2018 Apr;32(4):387-398. doi: 10.1007/s40263-018-0498-4. PMID 29532440

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 77 subjects with Parkinson's disease (PD) and Levodopa-induced Dyskinesia (LID) were randomized at 32 study sites in the United States, Germany, France, Spain, and Austria. The first subject was randomized on 23 October 2014 and the last subject completed on 10 March 2016.
Pre-assignment Details: All randomized subjects who received ≥ 1 dose of study drug and provided ≥ 1 postbaseline efficacy assessment (75) were included in both the Safety Analysis Population and the Modified Intent-to-Treat (MITT) population (with 38 subjects in the placebo group and 37 in the ADS-5102 group).
Groups:
- Placebo: Placebo: oral capsules administered once nightly at bedtime for 13 weeks
- ADS-5102 (Amantadine HCl Extended Release): 340 mg dose of ADS-5102 (amantadine hydrochloride [HCl] extended release): oral capsules administered once nightly at bedtime for 13 weeks
Period: Overall Study
Arm/Group | Placebo | ADS-5102 (Amantadine HCl Extended Release)
Started | 39 | 38
Received Study Drug | 38 | 37
Completed | 35 | 29
Not Completed | 4 | 9
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Did Not Receive Study Drug | 1 | 1
Not completed — Subject Unwilling to Proceed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Population
Groups:
- ADS-5102 (Amantadine HCl Extended Release): 340 mg dose of ADS-5102 (amantadine HCl extended release): oral capsules administered once nightly at bedtime for 13 weeks
- Total: Total of all reporting groups
Arm/Group | Placebo | ADS-5102 (Amantadine HCl Extended Release) | Total
Number analyzed (Participants) | 38 | 37 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 16 | 31
  >=65 years | 23 | 21 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (9.08) | 64.7 (9.66) | 64.8 (9.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 20 | 19 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 5 | 5
  Not Hispanic or Latino | 38 | 32 | 70
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 38 | 36 | 74
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 15 | 23
  Europe | 30 | 22 | 52
Unified Dyskinesia Rating Scale (UDysRS) [Mean (Standard Deviation); unit: units on a scale] — The UDysRS is a dyskinesia rating scale that evaluates involuntary movements associated with PD; the UDysRS consists of the following sub-parts: IA, IB, IIA, IIB, III, and IV. The total score is the sum of all individual sub-parts, and scores for this measure can range from 0-104. The total objective score is the sum of Part III (which measures objective impairment) and Part IV (which measures objective disability), and scores for this measure can range from 0-44. For both the total score and total objective score, a higher score indicates more severe PD.
  units on a scale
    Total Score | 41.2 (10.32) | 40.2 (13.06) | 40.7 (11.68)
    Total Objective Score (Parts III, IV) | 15.9 (7.00) | 18.1 (7.99) | 17.0 (7.53)
PD Home Diary [Mean (Standard Deviation); unit: hours] — A PD home diary was used to score 5 different conditions in 30-minute intervals: ASLEEP, OFF, ON (ie, had adequate control of PD symptoms) without dyskinesia, ON with non-troublesome dyskinesia, and ON with troublesome dyskinesia.
  Total time with dyskinesia includes ON time with non-troublesome and troublesome dyskinesia.
  hours
    ON time without troublesome dyskinesia | 7.79 (3.249) | 8.77 (2.457) | 8.27 (2.909)
    ON time with troublesome dyskinesia | 6.02 (3.353) | 4.71 (2.509) | 5.37 (3.020)
    OFF time | 1.98 (1.687) | 2.62 (2.015) | 2.30 (1.871)
    Asleep time | 8.21 (1.643) | 7.91 (1.502) | 8.06 (1.572)
Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) [Mean (Standard Deviation); unit: units on a scale] — The MDS-UPDRS Parts I, II, III, and IV examined non-motor experiences of daily living, motor experiences of daily living, motor examination, and motor complications, respectively. Each Part contains items/questions, each rated on a scale from 0 (normal) to 4 (severe). The range of total scores for each Part is as follows: Part I, 0-52; Part II, 0-52; Part III, 0-132; Part IV, 0-24. Combined Parts I, II, and III is the sum of scores from Parts I, II, and III and has a scale range of 0-236. Parts 4.1 and 4.2 each has a scale range of 0-4. Higher scores indicate more severe PD.
  units on a scale
    Part I | 9.9 (4.86) | 11.3 (5.87) | 10.6 (5.39)
    Part II | 14.8 (6.06) | 14.1 (6.15) | 14.4 (6.07)
    Part III | 21.4 (10.22) | 21.2 (9.24) | 21.3 (9.68)
    Combined Parts I, II, and III | 46.1 (17.00) | 46.6 (14.76) | 46.3 (15.83)
    Part IV | 11.1 (2.40) | 9.8 (2.78) | 10.5 (2.66)
    Part IV, Item 4.1 | 2.8 (0.94) | 2.2 (0.81) | 2.5 (0.92)
    Part IV, Item 4.2 | 2.5 (0.51) | 2.5 (0.61) | 2.5 (0.55)
Time Since PD Diagnosis [Mean (Standard Deviation); unit: years] | 10.71 (4.265) | 10.40 (5.105) | 10.55 (4.669)
Duration of Levodopa Treatment [Mean (Standard Deviation); unit: years] | 8.54 (4.845) | 7.69 (4.121) | 8.12 (4.493)
Duration of LID [Mean (Standard Deviation); unit: years] | 3.98 (2.566) | 3.78 (3.160) | 3.88 (2.857)
Hoehn and Yahr Stage [Mean (Standard Deviation); unit: units on a scale] — The Hoehn and Yahr scale, from 1-5, describes the subject's PD progression. The higher the score the more severe the symptoms of PD.
  units on a scale | 2.4 (0.55) | 2.1 (0.60) | 2.2 (0.59)
Subjects taking Antiparkinson Medication [Count of Participants; unit: Participants] — Subjects may have been taking more than 1 antiparkinson medication at Baseline.
  Participants
    Levodopa | 38 | 37 | 75
    Dopamine Agonists | 25 | 21 | 46
    MAO Inhibitors | 20 | 17 | 37
    COMT Inhibitors | 1 | 3 | 4
    Anticholinergics | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in the Unified Dyskinesia Rating Scale (UDysRS) Total Score
Description: The UDysRS is a dyskinesia rating scale from 0-104; it evaluates involuntary movements associated with PD. A higher score indicates more severe PD. The UDysRS was measured at Baseline and Weeks 2, 4, 8, and 12.
Time Frame: Baseline to Week 12
Population: MITT population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | ADS-5102 (Amantadine HCl Extended Release)
Number analyzed (Participants) | 38 | 37
units on a scale | -6.3 (2.08) | -20.7 (2.20)
Statistical Analysis 1: Comparison: ADS-5102 (Amantadine HCl Extended Release); 32 subjects per treatment arm provided 90% power using a 2-sided test at 5% significance; Test type: Superiority; p < 0.0001, Linear Mixed Model w/ Repeated Measures; Change from baseline is a dependent variable; the baseline value is a continuous covariate; Least Squares Mean Difference = -14.4, 95% CI 2-sided [-20.4 to -8.3], Standard Error of Mean 3.03

2. Secondary Outcome: Change in the Standardized PD Home Diary (ON Time Without Dyskinesia, ON Time With Troublesome Dyskinesia, OFF Time)
Description: A PD home diary was used to score 5 different conditions in 30-minute intervals: ASLEEP, OFF, ON (ie, had adequate control of PD symptoms) without dyskinesia, ON with non-troublesome dyskinesia, and ON with troublesome dyskinesia. The results were based on 2 consecutive 24-hour diaries taken prior to the day of randomization and prior to the Week 2, 4, 8, and 12 visits.
Time Frame: Baseline to Week 12
Population: MITT population
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Placebo | ADS-5102 (Amantadine HCl Extended Release)
Number analyzed (Participants) | 38 | 37
hours
  Change in ON time without troublesome dyskinesia | 2.05 (0.526) | 3.95 (0.562)
  Change in ON time with troublesome dyskinesia | -2.47 (0.436) | -3.61 (0.468)
  Change in OFF time | 0.61 (0.313) | -0.49 (0.336)
Statistical Analysis 1: Comparison: ADS-5102 (Amantadine HCl Extended Release); Test type: Superiority; p = 0.0168, Linear Mixed Model w/ Repeated Measures — Change from Baseline in ON time without troublesome dyskinesia; Least Squares Mean Difference = 1.90, 95% CI 2-sided [0.35 to 3.45], Standard Error of Mean 0.775
Statistical Analysis 2: Comparison: ADS-5102 (Amantadine HCl Extended Release); Test type: Superiority; p = 0.0853, Linear Mixed Model w/ Repeated Measures — Change from Baseline in ON time with troublesome dyskinesia; Least Squares Mean Difference = -1.13, 95% CI 2-sided [-2.42 to 0.16], Standard Error of Mean 0.648
Statistical Analysis 3: Comparison: ADS-5102 (Amantadine HCl Extended Release); Test type: Superiority; p = 0.0199, Linear Mixed Model w/ Repeated Measures — Change from Baseline in OFF time; Least Squares Mean Difference = -1.10, 95% CI 2-sided [-2.02 to -0.18], Standard Error of Mean 0.461

ADVERSE EVENTS:
Time Frame: Baseline through Week 13
Arm/Group | Placebo | ADS-5102 (Amantadine HCl Extended Release)
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/38 | 4/37
Other Adverse Events (participants affected / at risk) | 19/38 | 31/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=38) | ADS-5102 (Amantadine HCl Extended Release) (N=37)
Suicide attempt (Psychiatric disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=38) | ADS-5102 (Amantadine HCl Extended Release) (N=37)
Dry mouth (Gastrointestinal disorders) | 1 | 5
Nausea (Gastrointestinal disorders) | 1 | 5
Decreased appetite (Metabolism and nutrition disorders) | 0 | 4
Insomnia (Psychiatric disorders) | 0 | 4
Orthostatic hypotension (Vascular disorders) | 0 | 4
Constipation (Gastrointestinal disorders) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 3
Hallucination (Pooled) (Psychiatric disorders) | 2 | 3 — consisted of auditory (0/38 in placebo, 1/37 in ADS-5102) and visual (2/38 in placebo, 3/37 in ADS-5102)
Apathy (Psychiatric disorders) | 0 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Depressed mood (Psychiatric disorders) | 0 | 2
Dizziness (Nervous system disorders) | 1 | 2
Dystonia (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 1 | 2
Malaise (General disorders) | 0 | 2
Somnolence (Nervous system disorders) | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Asthenia (General disorders) | 2 | 1
Nasopharyngitis (Infections and infestations) | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Affect lability (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Middle insomnia (Psychiatric disorders) | 0 | 1
Nervousness (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0
Freezing phenomenon (Nervous system disorders) | 0 | 1
Intracranial venous sinus thrombosis (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 1
Transverse sinus thrombosis (Nervous system disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Peripheral coldness (Vascular disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Hunger (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Nocturia (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 1
Photophobia (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 1
Vitreous floaters (Eye disorders) | 1 | 0
Visual impairement (Eye disorders) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Weight increased (Investigations) | 0 | 1
Glomerular filtration rate decreased (Investigations) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No